CLINICAL TRIAL: NCT00799916
Title: Saline Solution Versus Voluven®: A Controlled Study of Fluid Resuscitation in Severe Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de La Plata (Other)
Collaborators: Clínica Bazterrica (Other); Sanatorio Otamendi y Miroli (Unknown); National Agency for Scientific and Technological Promotion, Argentina (Other)
Responsible Party: Analía Pérez/Dirección de evaluación de medicamentos, Administración Nacional de Medicamentos, Alimentos y Tecnología Médica (ANMAT)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM 001
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Sepsis
Keywords: Sepsis; Fluid resuscitation; Voluven; Colloids; Saline solution; Crystalloids; Sublingual microcirculation
MeSH Terms: conditions — Sepsis | interventions — Resuscitation; HES 130-0.4; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voluven (Active Comparator): Resuscitation fluid: Voluven (R)
  Interventions: Drug: Resuscitation (Voluven)
- Saline (Active Comparator): Resuscitation fluid: Saline solution
  Interventions: Drug: Resuscitation (Saline)

INTERVENTIONS:
Drug: Resuscitation (Voluven) — Resuscitation aimed at venous oxygen saturation higher than 70%
  Arms: Voluven
Drug: Resuscitation (Saline) — Resuscitation aimed at venous oxygen saturation higher than 70%
  Arms: Saline

SUMMARY:
Fluid resuscitation of severe sepsis may consist of natural or artificial colloids or crystalloids. There is no evidence-based support for one type of fluid over another.

The investigators hypothesis is that fluid resuscitation with Voluven® is advantageous to normal saline solution to improve sublingual microcirculation.

DETAILED DESCRIPTION:
Shock is the failure of circulatory system to maintain adequate cellular perfusion. Septic shock is primarily a form of distributive shock and is characterized by ineffective tissue oxygen delivery and extraction associated with inappropriate peripheral vasodilation despite preserved or increased cardiac output. In sepsis, a complex interaction between pathologic vasodilation, relative and absolute hypovolemia, myocardial dysfunction, and altered blood flow distribution occurs due to the inflammatory response to infection. Even after the restoration of intravascular volume, microcirculatory abnormalities may persist and lead to maldistribution of cardiac output.

Notwithstanding the complexity of its pathophysiology and treatment, to maintain adequate organ perfusion is a main goal in the management of severe sepsis and septic shock. For this purpose, optimization of intravascular volume and preload is the more important step. Fluid challenge is a term used to describe the initial volume expansion period in which the response of the patient to fluid administration is carefully evaluated. During this process, large amounts of fluids may be administered over a short period of time under close monitoring to evaluate the patient's response and avoid the development of pulmonary edema. Fluid challenge should be given in all patients suspected of hypovolemia. Fluid resuscitation may consist of natural or artificial colloids or crystalloids. There is no evidence-based support for one type of fluid over another. As the volume of distribution is much larger for crystalloids than for colloids, resuscitation with crystalloids requires more fluid to achieve the same end points and might result in more edema. In addition, post-hoc analysis and experimental studies suggest that colloids might be superior to crystalloids, in terms of physiologic end-points, recruitment of the microcirculation and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis

Exclusion Criteria:

* Age of less than 18 years
* Pregnancy, or the presence of an acute cerebral vascular event, acute coronary syndrome, acute pulmonary edema, status asthmatics
* Cardiac dysrhythmias (as a primary diagnosis), contraindication to central venous catheterization, active gastrointestinal hemorrhage, seizure
* Drug overdose, burn injury, trauma, a requirement for immediate surgery, uncured cancer (during chemotherapy
* Immunosuppression (because of organ transplantation or systemic disease), do-not-resuscitate status, advanced directives restricting implementation of the protocol
* Delayed admission to ICU from emergency department (more than 4 hours), or fluid resuscitation previous to ICU with more than 1,500 cc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Sublingual microcirculation | 24 hour

SECONDARY OUTCOMES:
Gases, hemoglobin and oxygen saturations | 24 hours
Electrolytes and lactate | 24 hours
Anion gap corrected to albumin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo Dubin, MD, Principal Investigator — Sanatorio Otamendi y Miroli
Locations (3):
- Argentina (3):
  - Clinica Bazterrica, Buenos Aires
  - Clínica Santa Isabel, Buenos Aires
  - Sanatorio Otamendi y Miroli, Buenos Aires

REFERENCES:
- [Derived] Dubin A, Pozo MO, Casabella CA, Murias G, Palizas F Jr, Moseinco MC, Kanoore Edul VS, Palizas F, Estenssoro E, Ince C. Comparison of 6% hydroxyethyl starch 130/0.4 and saline solution for resuscitation of the microcirculation during the early goal-directed therapy of septic patients. J Crit Care. 2010 Dec;25(4):659.e1-8. doi: 10.1016/j.jcrc.2010.04.007. Epub 2010 Sep 1. PMID 20813485